CLINICAL TRIAL: NCT05570175
Title: Effectiveness of Mobile Application Self-management Program (App) for Joint Protection and Physical Activity in Patients With Rheumatoid Arthritis
Brief Title: Effects of a Mobile Application RA Joint Protection and Activity Self-management Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ChangGungMHappRA
Record Dates: First submitted 2022-10-04; First posted 2022-10-06 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2022-10

CONDITIONS: Arthritis, Rheumatoid
Keywords: self-management, self-efficacy, mobile application
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to experimental group who received a mobile application RA joint protection and activity self-management program based on self-efficacy theory for 6 weeks, and a control group receiving standard rheumatology care only.
Who Masked: Outcomes Assessor
Masking Description: The researcher who collected the data and the researcher who applied the intervention program was never the same.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The intervention group received a mobile application RA joint protection and activity self-management program based on self-efficacy theory for 6 weeks.
  Interventions: Behavioral: Mobile application RA joint protection and activity self-management program
- control group (No Intervention): The control group received general information on rheumatoid arthritis care and follow-up.

INTERVENTIONS:
Behavioral: Mobile application RA joint protection and activity self-management program — The intervention group received a mobile application RA joint protection and activity self-management program based on self-efficacy theory for 6 weeks. The program was based on self-efficacy theory and proposes that self-efficacy is influenced by four information sources: mastery of experience, social modeling, social persuasion and one's physical and emotional states. To enhance participants' self-management skill, the following strategies were employed: peer story-telling, assessment, family involvement, goal setting, self-monitoring, self-evaluation, and phone calls consultation.
  Arms: intervention group

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of mobile application self-management program (App) for joint protection and physical activity in patients with rheumatoid arthritis. Intervention group received an app self-management program. The researchers compared the effects of the experimental group and the control group in disease activity, physical functioning, self-efficacy, depression, and self-management behavior.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a persistent systemic disease. World Health Organization commented that a crucial goal of heath care for RA is prevention of loss of daily function by patients' self-management (SM) skills; however, the evidences from literature presented that there are some limitations in traditional self-management interventions, and a comprehensive rheumatoid arthritis online self-management program for RA patients' day-to-day self-managing is limited in Taiwan. The goal of this clinical trial is to evaluate the effectiveness of mobile application self-management program (App) for joint protection and physical activity in patients with rheumatoid arthritis. The project was designed to implement and evaluate the app rheumatoid arthritis self-management program for RA patients using two groups experimental design. A medical center in northern Taiwan was selected and patients who visited the RA departments were eligible for the study if they are diagnosis of RA, age of 20 years or over, disease considered by the treating rheumatologist to have been stable for at least 12 weeks, able to communicate with researcher, and use a mobile. Patients were excluded if they are suffering from other terminal illnesses, severe dementia or another debilitating psychiatric disorder, or living in a long-term care facility. After completion of baseline data, patients were randomly allocated to the intervention or control group using a computerized allocation procedure and follow the CONSORT flow diagram. Control patients received usual care, and the intervention group received the 6-week app rheumatoid arthritis self-management program which based on self-efficacy theory. The independent variable of the program was the four information include mastery experience, social modeling, social persuasion and physical and emotional states, and the strategies involve education, goal setting and attainment, self-monitoring, and phone calls. All participants were followed up for 6 months, and the data were collected at the baseline, 8, and 12 weeks. The statistics with the generalized estimating equation analysis was used to evaluate the outcomes such as the disease activity (DAS-28), arthritis self-efficacy (ASE), physical functioning (MHAQ), depression, and self-management behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with RA
* Age of 20 years or over
* Disease considered have been stable for at least 3 months
* Able to understand and comply with the study treatment
* Use a mobile

Exclusion Criteria:

* Suffering from other terminal illnesses, severe dementia or another debilitating psychiatric disorder
* Living in a long-term care facility

Min Age: 20 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Su-Hui Chen, PhD, Principal Investigator — Professor, School of Nursing, Chang Gung University of Science and Technology
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

REFERENCES:
- [Derived] Shao JH, Yu KH, Kao YC, Liang YC, Chen SH. Effects of a Smartphone App-Based Intervention on Rheumatoid Arthritis Self-Management Efficacy: A Randomized Controlled Trial. J Nurs Res. 2024 Oct 1;32(5):e349. doi: 10.1097/jnr.0000000000000638. PMID 39514777

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 25 | 21
Completed | 21 | 21
Not Completed | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 25 | 21 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.84 (10.54) | 62.1 (16.86) | 58.70 (13.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 17 | 39
  Male | 3 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 25 | 21 | 46
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 25 | 21 | 46
Duration of RA [Mean (Standard Deviation); unit: years] | 9.06 (5.33) | 14.33 (12.12) | 11.47 (9.35)

OUTCOME MEASURES:

1. Primary Outcome: Self-management Behaviors
Description: To assess self-management behaviors the researchers developed a joint activity and protection self-management behaviors scale. The scale consists of eight items and ranges from zero for 'never' to four for 'always'. The range of the score will be 0-32, higher scores indicate a better level of use of each of the self-management behavior.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 21
score on a scale | 13.24 (5.67) | 14.76 (6.71)

2. Secondary Outcome: Disease Activity
Description: Disease activity was measured using the DAS-28 (Disease Activity Score-28) which evaluated 28 tender and swollen joint counts of rheumatoid arthritis patients. This scale was used to calculate the 28 tender and swollen joint counts. Scores can range from 0 to 9.4. The lower score represent a better RA outcome.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 21
score on a scale | 3.45 (1.23) | 3.57 (0.81)

3. Secondary Outcome: Arthritis Self-efficacy- Pain
Description: We used the arthritis self-efficacy-pain (ASE-pain) to measure RA patients' pain self-efficacy. The ASE-pain used visual analogue scales (0-10), in which 0 means 'very uncertain' and 10 means 'very certain'; a higher score refers to better self-efficacy. This scale have 5 items, therefore, the score range will be 0-50.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 21
score on a scale | 24.08 (13.47) | 24.38 (16.63)

4. Secondary Outcome: Arthritis Self-efficacy- Other
Description: We used the arthritis self-efficacy-other (ASE-OS) to measure RA patients' other symptoms self-efficacy. The ASE-OS used visual analogue scales (0-10), in which 0 means 'very uncertain' and 10 means 'very certain'; a higher score refers to better self-efficacy. This scale have 6 items, therefore, the score range will be 0-60.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 21
score on a scale | 30.48 (15.75) | 33.00 (16.51)

5. Secondary Outcome: Physical Functioning
Description: The 8-item Modified Health Assessment Questionnaire (MHAQ) was used to measure the physical functioning for this study. The MHAQ measures eight activities such as dressing and grooming, arising, eating, walking, hygiene, reach grip, and common daily activities. Items are rated from 1 = without difficulty, to 4 = unable to do; a lower score indicates a better ability to conduct daily activities. The range of the score will be 8-32.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 21
score on a scale | 23.32 (4.34) | 23.10 (2.97)

ADVERSE EVENTS:
Time Frame: All-cause mortality, serious, and other adverse events were not monitored/assessed.
Description: 0
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT05570175/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT05570175/SAP_001.pdf